CLINICAL TRIAL: NCT05084066
Title: A Study on the Phenomenon of Remote Ischaemic Preconditioning in Patients With Peripheral Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tartu University Hospital (Other)
Responsible Party: Principal Investigator, Jaak Kals, Professor, University of Tartu
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 21082
Record Dates: First submitted 2021-09-21; First posted 2021-10-19 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Peripheral Arterial Disease
Keywords: Intermittent Claudication; Total Walking Distance; Initial Claudication Distance; Time to Relief of Claudication; Arterial Stiffness; VASCUQOL-6; Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): 20 patients with PAD and claudication
  Interventions: Other: Repeated remote ischemic preconditioning
- Control group (sham) (Sham Comparator): 20 patients with PAD and claudication
  Interventions: Other: Simulation of repeated remote ischemic preconditioning (sham)

INTERVENTIONS:
Other: Repeated remote ischemic preconditioning — An automated device performs four 5-minute episodes of upper limb ischemia in which the cuff pressure in the experimental group remains at 200 mmHg for 5 minutes, causing and ensuring ischemia. Ischemic episodes alternate with 5-minute reperfusion. The intervention lasts a total of 35 minutes. The participant places the device on his upper arm and presses the "Start" button, starting the intervention. The intervention takes place at rest in the patient's home environment daily for 28 days. During the first visit to the research center, the research assistant teaches the participant how to use the device. The device measures the patient's blood pressure at the start of the intervention. If the patient's blood pressure is above 200 mmHg, the device will not perform the intervention.
  Arms: Experimental group
Other: Simulation of repeated remote ischemic preconditioning (sham) — The automated device simulates the intervention of the experimental group with the difference that the device does not apply pressure to the upper limb and, therefore, no ischemia occurs.
  Arms: Control group (sham)

SUMMARY:
This study aims to evaluate whether remote ischemic preconditioning (RIPC) daily for 28 days reduces the symptoms of intermittent claudication in patients with peripheral artery disease (PAD). The study evaluates the effect of RIPC on patients' total walking distance (TWC), initial claudication distance (ICD), and time to relief of claudication (TRC). In addition, the trial investigates the effect of RIPC on different arterial functional characteristics and low molecular weight metabolites in serum and affected skeletal muscle.

DETAILED DESCRIPTION:
A research hypothesis is that repeated remote ischemic preconditioning (RIPC) daily for 28 days reduces the symptoms of intermittent claudication in patients with peripheral artery disease (PAD).

The investigators plan to conduct a randomized controlled trial. Clinically stable patients with PAD and intermittent claudication are randomly allocated to receive a repeated RIPC or sham for 28 days. An automated device generates RIPC. One cycle of RIPC consists of 4 cycles of 5-min upper limb ischemia followed by 5-min reperfusion (lasting a total of 35 minutes). The participant places the device on his upper arm and presses the "Start "button, starting the intervention. The intervention occurs at rest in the participant's home environment. The first intervention takes place in the research center, where the research assistant teaches the participant how to use the device. In the sham group, a RIPC imitation is performed. The sham device has the same sound and light effects as the active device; the only difference is that the pressure in the cuff does not increase, so ischemia does not occur.

Randomization is performed using blocks. Each block has 2-4 subjects. Subjects are divided according to smoking status (active smoker yes/no) and age (≥ 65 years or < 65 years old). Randomized letters (whether the subject will go into the experimental group or the sham group) are placed in opaque envelopes, which are opened right before the first intervention.

Participants will visit the research center twice. During the first visit, they fill in the VASCUQOL-6 questionnaire to evaluate their symptoms and health-related quality of life. In addition, the investigators collect participants' blood and urine samples, measure their arterial stiffness parameters and assess symptom-free and maximal walking distance on a treadmill. The investigators will take a skeletal muscle biopsy from the first ten participants in each group using a tiny percutaneous needle biopsy (TPNB) technique to measure low molecular weight metabolites in affected skeletal muscle.

These steps are repeated on the second visit (after 28 days of intervention). After data collection is completed, a statistical analysis is performed to evaluate whether RIPC improves participants' maximal walking distance, arterial stiffness, and metabolic parameters.

ELIGIBILITY:
Inclusion Criteria:

* Peripheral arterial disease, which causes claudication
* Patients who have given written informed consent and are undergoing conservative treatment for claudication (continuous treatment for at least three months)
* Patients with lower limb atherosclerosis Fontaine class IIA or IIB
* The primary limiter of walking is claudication, not any other condition
* Ankle-brachial index (ABI) ≤ 0,9 in symptomatic lower limb

Exclusion Criteria:

* Female gender
* Resting blood pressure > 200 mmHg
* Fontaine class III or IV
* eGFR < 30 ml/min/1,73 m2
* Home oxygen therapy or severe COPD (GOLD 3-4)
* Heart failure NYHA III-IV
* Stable angina pectoris
* Clinically severe COVID-19 infection in the last three months
* History of malignancy (within the last five years)
* Persistent or permanent atrial fibrillation or flutter
* Acute myocardial infarction in the last three months
* Residual signs of cerebral infarction that impede movement
* Significant atherosclerosis of peripheral arteries of the upper limb (symptomatic)
* History of deep vein thrombosis of the upper limb
* Diabetic polyneuropathy
* Under 18 years of age
* Patients who are unable to follow the study regimen

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-04-18 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Total Walking Distance at 28 Days | 28 days
  Maximal walking distance performed on a treadmill test

SECONDARY OUTCOMES:
Change from Baseline Initial Claudication Distance at 28 Days | 28 days
  The distance walked at the onset of claudication pain (assessed on a treadmill test)
Change from Baseline Time to Relief of Claudication at 28 Days | 28 days
  The amount of time it takes for the pain to go away after patient stops walking (assessed with stopwatch)
Change from Baseline Carotid-Femoral Pulse Wave Velocity at 28 Days | 28 days
  A measure of arterial stiffness (measured with SphygmoCor XCEL 7.0)
Change from Baseline Augmentation Index at 28 Days | 28 days
  A parameter of arterial stiffness (measured with SphygmoCor XCEL 7.0)
Change from Baseline Low Molecular Weight Metabolite Levels in Serum at 28 Days | 28 days
  A variety of acylcarnitines, amino acids, biogenic amines, glycerophospholipids, sphingolipids, and sugars measured using AbsoluteIDQ® p180 kit
Change from Baseline Low Molecular Weight Metabolite Levels in Muscle Biopsy Specimen at 28 Days | 28 days
  A variety of acylcarnitines, amino acids, biogenic amines, glycerophospholipids, sphingolipids, and sugars measured using AbsoluteIDQ® p180 kit
Change from Baseline Health-Related Quality of Life in PAD at 28 Days | 28 days
  Measured with Vascular Quality of Life Questionnaire-6 (VASCUQOL-6 questionnaire). The questionnaire consists of six questions. Every question has a 4-point response scale. An overall score ranges from 6 (worst) to 24 (best health-related quality of life) when summarizing the points.
Incidence of Major Adverse Cardiovascular Events (MACE) One Year after the Intervention | One year after the intervention
  Incidence of myocardial infarction, stroke, hospitalization because of heart failure and revascularization, including percutaneous coronary intervention and coronary artery bypass graft one year after the intervention
Incidence of Major Limb Events (MALE) One Year after the Intervention | One year after the intervention
  Incidence of acute limb ischemia, including thrombectomy and thrombolysis, major amputation at or above the ankle, or need for surgical peripheral revascularization one year after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jaak Kals, PhD, Principal Investigator — University of Tartu
Locations (1):
- Tartu University Hospital, Tartu, Estonia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eerik K, Kasepalu T, Post H, Eha J, Kals M, Bjorck M, Kals J. Effects of Repeated Remote Ischaemic Preconditioning on Arterial Stiffness, Organ Damage, and Oxidative Stress in Patients with Intermittent Claudication: A Sham Controlled Randomised Trial. Eur J Vasc Endovasc Surg. 2025 Jun 24:S1078-5884(25)00575-1. doi: 10.1016/j.ejvs.2025.06.046. Online ahead of print. PMID 40571146
- [Derived] Eerik K, Kasepalu T, Post H, Eha J, Kals M, Kals J. Editor's Choice - Daily Remote Ischaemic Preconditioning for Intermittent Claudication: A Sham Controlled Randomised Trial. Eur J Vasc Endovasc Surg. 2025 Feb;69(2):295-302. doi: 10.1016/j.ejvs.2024.10.047. Epub 2024 Nov 8. PMID 39522584